CLINICAL TRIAL: NCT03702972
Title: Contribution of Thermal Imaging in Determining the Depth of Pediatric Acute Burns: a Prospective Observational Study
Brief Title: Thermal Imaging and Pediatric Burns
Acronym: FLIRPED
Status: Withdrawn | Type: Observational
Why Stopped: Essential equipment unavailable
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18021J; 2018-A01154-51 (Other: ANSM)
Record Dates: First submitted 2018-09-28; First posted 2018-10-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2018-08

CONDITIONS: Burns Second Degree
Keywords: Burn; Pediatry; Flir One Thermal Imager; Depth determination
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The need to cover a burn with a skin graft is determined primarily by its depth. In fact only burns of the second deep degree or the third degree are likely to be grafted. However, if the diagnosis is obvious in the case of third degree burns, second degree burns are often "mixed" with more or less deep areas, especially in pediatrics.

Clinical experience and daily observation of the burn since its occurrence currently determine the indication for surgery. In practice, it is rare to be able to determine with certainty whether a second degree mixed burn will require a graft before the 10-12th day of evolution. There are currently devices that can help refine the diagnosis such as laser Doppler, but they are expensive devices, and not 100% reliable. The thermal camera Flir-one® attaches to a smartphone or tablet and allows thanks to a free application, to obtain a thermogram of the pointed area. This is a device used to detect insulation deficits in the building sector. Knowing that a deep burn, by devascularization, will have an external temperature lower than a superficial burn, a thermogram would thus make it possible to better identify the deep zones and the superficial zones of the burn. One study showed a good sensitivity and specificity of the device but it was a population of adult patients. This determined that a difference in skin temperature between a deep burned area and healthy skin should be at least 1.15 ° C in favor of healthy skin, to retain a burn as deep, and not to operate so-called superficial burn if this difference was below this threshold. However, further studies would be needed to demonstrate the validity of this method in clinical practice.

DETAILED DESCRIPTION:
All patients under 18, with acute burns (<10 days of development), surface area <10%, second degree, hospitalized from 22/01/18 in the plastic surgery department and burns Trousseau Hospital in Paris, subject to the non-opposition of parental authority. 500000 pediatric burns are counted each year in France. In 2005, they resulted in 5109 hospital stays 2. Improving the accuracy of the diagnosis before 10 days of evolution would make it possible to graft the children who needed it more quickly and thus shorten the length of hospital stay. It is therefore a public health issue, with a significant medical and economic impact.

Description of the item (s) being researched

It involves collecting, through a thermal camera, a temperature difference between a second-degree burn zone and an adjacent healthy zone, in order to prove that this difference, can make it possible to retain the burn as deep, and can therefore guide a surgical decision.

Justification of the duration of the research.

According to the same study in adults1, the number of patients to be included was 41 to obtain sufficient power for a statistical analysis of the same data collected in this study, and according to the same methodology. A duration of 4 months seems compatible with such recruitment in the specialized center for treating pediatric burns at the Trousseau Hospital in Paris.

Goal of the study: Objectively determine the depth of pediatric acute burns using a thermal imaging camera.

METHOD AND POPULATION

Main evaluation criterion Measurement of Δ T = temperature difference between the burned area and an adjacent healthy area of 3cm, or contralateral if extremity burns, with the thermal camera, by a blind surgeon the final evaluation of the depth (between D10 and D14 ).

The thermograms will be read at three different times, from the moment of admission to hospital or after the patient has been cured by:

* T1: D1 to D4 of the burn
* T2: D4 to D7 of the burn
* T3: D7 to D10 of the burn.

Secondary evaluation criteria Interest of the repeated measurements to determine if the evolution of ΔT is also an index reflecting the depth of the burn.

Recruitment of the population Hospitalized patients from 22/01/18 in the Pediatric Burn Surgery Department of Trousseau Hospital in Paris.

Eligibility criteria (inclusion and non-inclusion criteria) Inclusion criteria: All patients <18 years of age, with acute burns (<10 days of progression) of the second degree of body surface area burned <10%, hospitalized from 22/01/18 in the plastic surgery department and burns at the Trousseau Hospital in Paris, subject to the non-opposition of parental authority.

Criteria for non-inclusion: First-degree burns, third-degree burns, fever episode not caused by burns, burn surgery before measurement, inability to communicate with the persons having parental authority.

Population monitoring Patients will be followed as usual as part of the nurse consultation consultation treatment every 2 days initially at the Trousseau Hospital Pediatric Burn Treatment Center, with surgical advice on how to proceed with care. local, as was already the case, then the pace will adapt to the pathology, with iterative appointments specialized consultation with the surgeon from 15 days after discharge and every 2 months until complete healing and definitive in the event of satisfactory evolution. In the case of surgery necessary for healing during hospitalization, the follow-up may last for a period of 2 years.

Risks AND VIGILANCE

Non-interventional research involving the human person presents no risk to patients.

The adverse effects observed in the patients participating in the research are notified by the investigators according to the local vigilance plans put in place as part of the care activities.

Terms of data collection

The collection of thermograms on thermal camera is performed by a blind surgeon of the operative decision of the burn. The thermograms will be read at three different times, from the moment of admission to hospital or after the patient has been cured by:

* T1: D1 to D4 of the burn
* T2: D4 to D7 of the burn
* T3: D7 to D10 of the burn

An operative decision or a continuation of the surgical care is recorded in the database at D10-14 in blind of the registered thermograms, by the only expertise of a surgeon different from that having measured the ΔT thus without modification of the care usually dispensed for each patient included.

The research does not foresee the use of data extracted from existing information systems or study bases already carried out.

Data circuit The collection of thermograms on a thermal camera is done by a surgeon who uses himself to transfer them by connectivity on the centralized computer database, protected, anonymized with a number given to each patient which only the surgeon having collected the thermograms knows the correspondence with the real identity. This surgeon does not participate in the operative decision of the patient and records it if necessary in the patient database after it is taken by the rest of the surgical team who remains blind thermograms and Δ T measured.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years,
* Acute burns (<10 days of evolution) of the second degree
* Body surface burned <10% of total body area
* Hospitalized patients for a period of 4 months and 15 days in the plastic surgery and burns department at Trousseau Hospital in Paris.
* Affiliates to the general system of social security as having the right of the holders of parental authority

Exclusion Criteria:

* Burns of the first degree,
* Third degree burns,
* fever episode not caused by burning,
* Surgical procedure on burn before measurement,
* Impossibility to communicate with the holders of the parental authority or opposition formulated to the participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minor patients hospitalized in the Burns Surgery Department at Trousseau Hospital with second degree burns less than 10 days old, less than 10% of total body surface area
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Temperature difference between burned zone and adjacent or contralateral healthy zone at time T3 | day 7 to day 10 from the day of the burn occurrence
  Δ T3 will be recorded from day 7 to day 10 once by the Flir One Thermal Imager

SECONDARY OUTCOMES:
Temperature difference between burned zone and adjacent or contralateral healthy zone at time s T1 | day 1 to day 4 from the day of the burn occurrence
  Δ T1 will be recorded from day 1 to day 4 once by the Flir One Thermal Imager
Temperature difference between burned zone and adjacent or contralateral healthy zone at time s T2 | day 4 to day 7 from the day of the burn occurrence
  Δ T2 will be recorded from day 4 to day 7 once by the Flir One Thermal Imager

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CASSIER, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No